CLINICAL TRIAL: NCT05105490
Title: PerQdisc PMCF1 Observational Trial to Evaluate the Clinical Performance and Safety of the PerQdisc Nucleus Replacement Device
Brief Title: Post Market Observational Trial for the PerQdisc Nucleus Replacement Device
Acronym: PMCF1
Status: Withdrawn | Type: Observational
Why Stopped: Study withdrawn upon CE mark receipt
Sponsor: Spinal Stabilization Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: PerQdisc PMCF1
Record Dates: First submitted 2021-10-11; First posted 2021-11-03 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Degenerative Disc Disease; Chronic Low-back Pain
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chronic Discogenic Low Back Pain: Patient is skeletally mature and between 21 and 60 years of age.
  Patient has Degenerative Disc Disease (DDD) at one or more levels
  between L1 and S1 but must have a single level identified as the pain generator.
  Patient has adequate disc height (6mm) at the level to be treated
  Patient is not responsive to conservative, non-surgical treatment for back pain.
  Interventions: Drug: PerQdisc

INTERVENTIONS:
Drug: PerQdisc — Observational trial to collect post-market safety and efficacy information in a limited number of human patients
  Other Names: PerQdisc Nucleus Replacement System

SUMMARY:
PerQdisc PMCF1 is a post-market clinical follow-up observational trial to follow subjects receiving a PerQdisc spinal implant for a duration of 5 years.

DETAILED DESCRIPTION:
This study will be a prospective, open-label, multi-center post-market observational study including 72 patients that will collect additional safety and efficacy data for the Spinal Stabilization Technologies PerQdisc Nucleus Replacement System. Primary endpoints will be used to assess the safety and efficacy of the PerQdisc device.

ELIGIBILITY:
Inclusion Criteria:

* Patient is skeletally mature and between 21 and 60 years of age.
* Patient has Degenerative Disc Disease (DDD) at one or more levels between L1 and S1 but must have a single level identified as the pain generator.
* Patient has adequate disc height (6mm) at the level to be treated
* Patient is not responsive to conservative, non-surgical treatment for back pain.
* Patient has signed the approved Informed Consent Form.

Exclusion Criteria:

* Patient has less than 6 mm of disc height.
* Patient has had prior lumbar spine surgery (nucleoplasty at non-index level is considered acceptable).
* Patient has had spinal fusion in the lumbar or thoracic intervertebral spaces. Cervical fusion is allowed as long as there are no neurologic deficits in the lower extremities.
* Patient has spondyloarthropathy or other spondylolisthesis greater than 2 mm.
* Patient has congenital moderate or severe spinal stenosis or epidural lipomatosis.
* Patient has significant facet disease. Significant is defined as pain improvement of 80% or more following image-guided medial branch blocks of the target level according to Spine Intervention Society (SIS) guidelines (diagnostic, contrast controlled).
* Patient has any known active malignancy.
* Patient has previously undergone or currently on immunosuppressive therapy. Steroids used to treat inflammation are allowed.
* Patient has active or local systemic infection.
* Patient has been diagnosed with hepatitis, rheumatoid arthritis, lupus erythematosus, or other autoimmune disease including Acquired Immune Deficiency Syndrome (AIDS), AIDS related Complex (ARC), and Human Immunodeficiency Virus (HIV).
* Patient has diabetes mellitus (Type 1 or 2) requiring daily insulin management.
* Patient has osteopenia of the spine (T-score of -1.0 or lower). A Bone Densiometry (DEXA) scan should be performed to rule out patients considered at risk for osteopenia.
* Patient has morbid obesity defined as a Body Mass Index (BMI) more than 40 or a weight of more than 45 kg (100 lbs.) over ideal body weight.
* Patient has a known allergy to silicone or barium sulfate.
* Patient has a significant disc herniation at the level to be treated. Significant is defined as a large extruded herniation that creates a risk for expulsion.
* Patient has a significant Schmorl's node in the level to be treated. Significant is defined as a large, rectangular or irregular shaped node that has an associated active inflammatory process (Modic I changes).
* Patient has motion of less than 3 degrees on pre-operative lateral flexion/extension radiographs.
* Protrusion of the 20A Imaging Balloon up to or beyond the outer margin of the vertebra during the imaging steps.
* Patient has a violated endplate as determined by imaging balloons during fluoroscopy.
* Patient has a disc space that is too narrow for implantation.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Skeletally mature patients, age 21-60 years, with chronic low back pain of discogenic origin that is non-responsive to conservative, non-surgical therapy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-12-31 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
PerQdisc Perfomance | 6 months post implant
  Change in Oswestry Disability Index (ODI) comparing baseline to follow up visits using a patient-reported outcome tool
PerQdisc Perfomance | 12 months post implant
  Change in Oswestry Disability Index (ODI) comparing baseline to follow up visits using a patient-reported outcome tool
PerQdisc Safety | 6 months post implant
  Incidence of device expulsion and device fracture following surgery based on follow up X-rays and MRI's
PerQdisc Safety | 12 months post implant
  Incidence of device expulsion and device fracture following surgery based on follow up x-rays and MRI's

SECONDARY OUTCOMES:
Incidence of Secondary Surgeries | 6 months, 12 months, and 5 years following surgery
  Incidence of revision surgery at the index level or other secondary lumbar surgery at a non-index level
Maintenance of Disc Height | 6 months, 12 months, and 5 years following surgery
  Intervertebral disc height (in mm) as measured on MRI post-surgery compared to baseline
Maintenance of Range of Motion | 6 months, 12 months, and 5 years following surgery
  Measurement of range of motion (expressed in degrees) at the index and adjacent levels at baseline compared to post-surgical follow-up using flexion/extension x-rays.
Maintenance of Neurologic Status | 6 months, 12 months, and 5 years following surgery
  Physical assessment evaluating nerve compression at baseline and post-surgical follow up using pain, motor strength, and sensation feedback from the patient on a 0 (no compression) to 5 (major compression) scale.
Use of Pain Medications | 6 months, 12 months, and 5 years following surgery
  Change in level of pain medication used comparing baseline to follow up visits based on a medication scale ranging from 0 to 4. 0 (no meds) to 4 (high dose opioids)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hess, MD, Study Director — Spinal Stabilization Technologies; Jeff Golan, MD, Study Director — Spinal Stabilization Technologies
Locations (1):
- Donauisar Klinikum Deggendorf, Deggendorf, Germany

IPD SHARING:
Plan to Share IPD: Yes
De-identified outcome data will be available to participating investigators
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available 1 year after the final patient has completed one-year follow-up. Additional data will be available after the final patient has completed 5 year follow up
Access Criteria: Data will be shared with investigators from a secure electronic database